CLINICAL TRIAL: NCT04793113
Title: A Study to Assess the Effects of Freshly Fit Meals on Body Weight and Wellness in Overweight and Obese Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Freshly, Inc. (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BIO-2105
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Low carbohydrate, high protein meals
  Interventions: Other: FreshlyFit Meals

INTERVENTIONS:
Other: FreshlyFit Meals — FreshlyFit meals are low carbohydrate, high protein meals

SUMMARY:
The primary objective of this trial is to examine the weight-loss efficacy of Freshly Fit meals, as well as body composition, waist/hip circumference, metabolic markers, and quality of life in overweight and obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 21-55 years of age, inclusive, at Visit 1 (Day -10).
* BMI of 25.00 to 34.99 kg/m2, inclusive, at Visits 1 and 2 (Day -10 and -3).
* Non-smoker and has no plans to change smoking habits during the study period.
* Willing to follow study instructions.
* Willing and able to comply with the visit schedule (e.g., subjects with travel plans and cannot fully comply with study instructions will be excluded).

Exclusion Criteria:

* Abnormal laboratory test result of clinical significance at Visit 1 (Day -10), at the discretion of the Investigator. One re-test will be allowed on a separate day prior to Visit 2 (Day -3) for subjects with abnormal laboratory test results.
* History or presence of clinically important cardiac, renal, hepatic, endocrine, pulmonary, biliary, pancreatic, or neurological disorders that may affect the subject's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Investigator.
* History of gastrointestinal surgery for weight reducing purposes.
* Participation in a weight loss trial within 12 mo of Visit 1 (Day -10).
* Weight loss or gain ≥10 lb (4.5 kg) within the 6 mo prior to Visit 1 (Day -10). Participation in a program/service intended to alter body weight (e.g., Nutrisystem, Weight Watchers, Noom) within 6 mo of Visit 1 (Day -10).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2021-09-23 (Estimated); Study Completion 2021-09-23 (Estimated)

PRIMARY OUTCOMES:
Weight Change | 16 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided